CLINICAL TRIAL: NCT04931498
Title: Molecular Investigation of GENetic Factors in Cardiovascular and Immune-related Traits and Diseases Using a BIOresource of Healthy Volunteers
Brief Title: Molecular Investigation of GENetic Factors in Cardiovascular and Immune-related Traits and Diseases Using a BIOresource of Healthy Volunteers (GENBIO)
Acronym: GENBIO
Status: Active, not recruiting | Type: Observational
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Principal Investigator, Dirk Paul, Principal Investigator, University of Cambridge
Other Study IDs: GENBIO
Record Dates: First submitted 2021-06-04; First posted 2021-06-18 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Cardiovascular Diseases
Keywords: Healthy Volunteers; Genetic Risk Markers for Disease; Coronary Heart Disease; Coronary Artery Disease; Immune Response; Red Blood Cells; Inflammation
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Coronary Artery Disease; Inflammation | interventions — Surveys and Questionnaires; Weights and Measures; Blood Pressure; Heart Rate; Blood Specimen Collection; GMP Reductase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- GMPR sub-study: Study population will be split into five haplotypes based on a combination of rare and common variants at the GMPR locus. A total of 26 volunteers per genotypic group in a comparison between heterozygous and homozygous individuals will be tested.
  Interventions: Other: Questionnaire; Other: Anthropometric measurements: height, weight, and body fat; Other: Blood pressure and heart rate; Procedure: Venepuncture (GMPR)
- SWAP70 sub-study: To assess genotype-specific effects on SWAP70 protein levels as well as coronary artery disease-related immune processes, we will recruit 50 volunteers stratified by variant genotype, i.e. major and minor homozygotes only (25 participants will be recruited to each group).
  Interventions: Other: Questionnaire; Other: Anthropometric measurements: height, weight, and body fat; Other: Blood pressure and heart rate; Procedure: Venepuncture (SWAP70)

INTERVENTIONS:
Other: Questionnaire — Medical history, demographics and lifestyle factors will be assessed by the participant.
Other: Anthropometric measurements: height, weight, and body fat — Height measured by stadiometer. Weight and body fat measured by Tanita scale bioelectrical impedance analysis.
Other: Blood pressure and heart rate — Parameters will be measured using a validated, automated device while seated and again after 3-5 min standing. All measurements will be done in triplicate.
Procedure: Venepuncture (GMPR) — A blood sample of approximately 50 ml of venous blood will be taken. From the obtained blood sample, measurements will include a full blood count and the following phenotyping tests:
  * Flow cytometry to quantify cell surface expression of key erythroid markers
  * Proteomic analysis of isolated erythrocytes using mass spectrometry
  Groups: GMPR sub-study
Procedure: Venepuncture (SWAP70) — A blood sample of approximately 50 ml of venous blood will be taken. From the obtained blood sample, measurements will include a full blood count and the following phenotyping tests:
  * Flow cytometry to quantify cell surface expression of key markers
  * Fluorescence-Activated Cell Sorting (FACS) to assess B-cell receptor signalling and to isolate cell type-specific RNA for transcriptome analysis
  * Immunoglobulin isotype titre analysis in plasma
  * Isolation of monocytes for subsequent use in phagocytosis assays
  Groups: SWAP70 sub-study

SUMMARY:
The risk of cardiovascular disease is determined by the complex interplay between an individual's genetic make-up, lifestyle, and the environment. The researchers in this observational, cross-sectional, recall-by-genotype study are investigating two potential genetic risk factors; the SWAP70 gene is thought to play a role in the immune response modulating cardiovascular disease risk and the GMPR gene plays a role in red blood cell formation. The investigators hope to identify and characterise distinct molecular and cellular mechanisms underlying candidate functional variants identified in genetic studies of cardiovascular and immune-related human traits and diseases.

Healthy volunteers who are part of the NIHR BioResource and have already been genotyped will be invited to the study based on their genotype of the candidate functional variants of interest. Volunteers will attend a single study visit, during which they will complete procedures including a medical, demographic and lifestyle factors questionnaire; height, weight and body fat assessments; in addition to blood pressure/heart rate measurements. A minimally invasive procedure of a venepuncture will be performed to assess the primary objectives of the study.

The obtained data may (1) improve understanding of biological and disease mechanisms; (2) identify potential drug targets; and (3) improve insight into the therapeutic potential and limitations of existing and emerging therapies.

This study is funded by the UK Medical Research Council, British Heart Foundation and NIHR Cambridge Biomedical Research Centre.

ELIGIBILITY:
Inclusion Criteria:

* Have consented to be part of the NIHR BioResource;
* Are aged 18 years and above;
* Have given written informed consent to participate in the GENBIO study;
* Are carriers or non-carriers of the candidate functional genetic variant(s) of interest.

Exclusion Criteria:

Have a chronic disease, including cardiovascular diseases, autoimmune diseases and cancer.

Additional exclusion criteria to be applied at the discretion/opinion of the CI/collaborator, based on the population of available volunteers for recall and the genetic variant of interest (e.g. allele frequency):

* Have a biological first-degree relatives (parents, brothers, sisters or children) who are suffering or have suffered from a disease/condition in the opinion of the CI/collaborator that, from a genetic standpoint, may affect the study validity;
* Are current regular smokers. Regular ex-smokers are suitable if they stopped smoking >10 years ago (regular defined as 1 pack year in both instances);
* Have ≥3 alcoholic drinks per day;
* Have a diagnosis of hypertension, or history of consistently high blood pressure readings, e.g. >140/90 mmHg;
* Have a diagnosis of hypercholesterolemia, or history of consistently high cholesterol levels, e.g. total cholesterol level >6 mmol/l;
* Are obese (i.e. BMI >30);
* Are unwilling to fast and not to consume products containing alcohol or caffeine 12 hours prior to procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will only recruit healthy volunteers who have previously consented to being contacted for future studies by the NIHR Cambridge BioResource, which is a panel of around 20,000 volunteers, both with and without health conditions, who are willing to be approached to participate in research studies investigating the links between genes, the environment, health and disease. Volunteers who join the NIHR BioResource have donated their DNA via a blood or saliva sample that is used together with other information, such as sex and ethnicity, to match them to specific research studies. Participants for this study are identified by having the appropriate genetic sequence in one of the two genetic loci we are investigating (SWAP70, GMPR).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Levels of GMPR protein in isolated erythrocytes | At baseline
  GMPR-specific measurement to be assessed by mass spectrometry, comparing results between different GMPR genotypic groups.
Levels of SWAP70 protein in immune cell subsets | At baseline
  SWAP70-specific measurement to be assessed by flow cytometry, comparing results between SWAP70 genotypic groups.
Proportion of immune cell types as measured using flow cytometric analysis | At baseline
  SWAP70-specific measurement to be assessed by flow cytometry (e.g. lymphoid and myeloid cell markers), comparing results between SWAP70 genotypic groups.
Levels of genes/transcripts in immune cell subsets | At baseline
  SWAP70-specific measurement to be assessed by RNA sequencing, comparing results between SWAP70 genotypic groups.
Concentration of immunoglobulin isotypes in plasma | At baseline
  SWAP70-specific measurement to be assessed by immunoglobulin isotype (IgM, IgG, IgA and IgE) analysis, comparing results SWAP70 genotypic groups.
Phagocytosis by monocytes as measured by colorimetric analysis (optical density) | At baseline
  SWAP70-specific measurement to be assessed by phagocytosis assays, comparing results between SWAP70 genotypic groups. The phagocytosis assay uses pre-labelled Zymosan particles as a pathogen for triggering phagocytosis. The engulfed Zymosan particles react with a specific substrate to produce a signal that can be detected by colorimetric analysis.

SECONDARY OUTCOMES:
Blood pressure (systolic and diastolic) | At baseline
  All study arms comparing results between genotypic groups.
Heart rate | At baseline
  All study arms comparing results between genotypic groups.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Paul, PhD, Principal Investigator — University of Cambridge
Locations (1):
- Department of Public Health and Primary Care, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Participant identifiable information is securely held, with restricted access, by the NIHR BioResource. Members of the research team carrying out the procedures will not be able to request the link to decode this information. Only the minimum required participant identifiable information (name and contact details) will be provided to the research team for the purpose of arranging study visits and completing the informed consent process. All research personnel will be sufficiently blinded of the genotype status of the healthy volunteers. All delegated research personnel that is responsible to conduct the data/statistical analysis will only analyse data that is anonymised of any patient identifiable data.